CLINICAL TRIAL: NCT05991284
Title: Sacubitril-Valsartan in Heart Failure With Preserved Ejection Fraction and Secondary Mitral Valve Regurgitation
Acronym: PRAISE-MR
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z-2023036
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Functional Mitral Regurgitation
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination; Standard of Care

STUDY DESIGN:
Intervention Model Description: Multicenter, Investigator-initiated, Prospective, Randomized trial with Open Blinded Endpoint
Who Masked: Outcomes Assessor
Masking Description: Blinded core echocardiography laboratory
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Active Comparator): Sacubitril-Valsartan (target dose 97/103 mg twice daily) on top of standard of care (including SGLT-2 inhibitor and MRA)
  Interventions: Drug: Sacubitril-valsartan; Drug: Standard of care
- Control arm (Placebo Comparator): Standard of care (including SGLT-2 inhibitor and MRA)
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Sacubitril-valsartan — sacubitril-valsartan (target dose 97/103 mg twice daily)
  Arms: Intervention arm
Drug: Standard of care — including SGLT-2 inhibitor and MRA

SUMMARY:
The main objective of this study is to assess the hemodynamic effects of sacubitril-valsartan in patients with heart failure with preserved ejection fraction and at least moderate atrial functional mitral regurgitation (AFMR), using a combination of cardiopulmonary exercise testing and stress echocardiography (referred to as CPETecho) at baseline and after six months of therapy. The patients included in this study will be randomly assigned to receive sacubitril-valsartan as an adjunct to standard medical care, as opposed to adhering solely to the standard of care which involves sodium-glucose cotransporter-2 (SGLT-2) inhibitor and mineralocorticoid receptor antagonist (MRA).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* New York Heart Association class II to IV.
* Written informed consent.
* Left ventricular (LV) ejection fraction ≥ 50%.
* Objective evidence of cardiac structural and/or functional abnormalities consistent with the presence of LV diastolic dysfunction/raised LV filling pressures, including raised natriuretic peptides.
* ≥ moderate functional MR assessed by transthoracic echocardiography within the previous year.

Exclusion Criteria:

* Systolic blood pressure < 100 mmHg.
* Potassium ≥ 5.2 mmol/L.
* Estimated Glomerular Filtration Rate ≤ 25 ml/min/1.73m².
* History of angioedema or unacceptable side effects during receipt of angiotensin converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARB).
* Structural mitral valve disease and previous or planned mitral valve intervention.
* Already receiving angiotensin receptor neprilysin inhibitor (ARNI, sacubitril-valsartan) therapy.
* Severe comorbid condition limiting life expectancy < 24 months or inability to perform a maximal CPETecho.
* Myocardial infarction, unstable angina, coronary revascularization within 12 weeks prior enrolment.
* Severe aortic, tricuspid or pulmonary valve disease.
* Pregnancy, lactation, or use of any method of contraception that is not highly effective.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean pulmonary arterial pressure over cardiac output slope assessed by CPETecho | Six months of treatment

SECONDARY OUTCOMES:
Change in peak oxygen uptake | Six months of treatment
Change in mitral effective regurgitant orifice area (EROA) | Six months of treatment
Change in natriuretic peptide levels | Six months of treatment
Change in left atrial volume (LAVI) | Six months of treatment
Change the minute ventilation over carbon dioxide production slope | Six months of treatment
Change in patient reported outcomes (Kansas City Cardiomyopathy Questionnaire, KCCQ-12) | Six months of treatment
Change in left atrial function (peak atrial longitudinal strain, PALS) | Six months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No